CLINICAL TRIAL: NCT07338708
Title: Assessment of Tolerance and Visual Outcomes After Bilateral Implantation of a Premium Type Intraocular Lens (Acrysof IQ Vivity IOL) in Patients With Cataract and Mild Keratoconus
Brief Title: Visual Outcomes and Quality of Life After Vivity EDOF IOL Implantation in Early-Stage Keratoconus
Acronym: VIVITY-KCONUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Emilio Pedrotti, Full Professor in Ophthalmology, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: prot. n. 22546
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cataract; Keratoconic Subjects
Keywords: EDOF IOL; Cataract; Vivity IOL; Early keratoconous; spectacle independence; optical quality; quality of life
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: This is a single-arm, prospective pilot study evaluating bilateral implantation of the AcrySof IQ Vivity Extended Depth of Focus (EDOF) intraocular lens (IOL) in patients with cataracts and early-stage, stable keratoconus. All participants receive the same intervention (Vivity EDOF IOL in both eyes, or its toric version if corneal astigmatism ≥1.00 D is present), with surgery on the second eye performed within 7 days of the first. There is no control or comparison group. The study explores whether this non-diffractive EDOF technology, which uses wavefront-shaping to extend focal range while preserving contrast sensitivity, can safely provide functional vision at multiple distances in a population (early keratoconus) traditionally considered unsuitable for premium IOLs due to corneal irregularities and higher-order aberrations. Outcomes are assessed at 3 months postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vivity EDOF IOL in Early Keratoconus (Experimental): Adults with cataracts and mild, stable bilateral keratoconus (ABCD stage 0-1) undergo bilateral implantation of the AcrySof IQ Vivity Extended Depth of Focus (EDOF) intraocular lens during standard phacoemulsification cataract surgery. The toric version is used in eyes with regular corneal astigmatism ≥1.00 D. Surgery is performed under topical anesthesia by the same surgeon, targeting bilateral emmetropia using Kane formula for IOL power calculation. The second eye is operated within 7 days of the first. The Vivity IOL is a non-diffractive EDOF lens utilizing X-WAVE wavefront-shaping technology to extend focal range without splitting light, designed to reduce visual disturbances while providing functional vision at distance, intermediate (66 cm), and near (40 cm). Comprehensive visual, optical quality, contrast sensitivity, and patient-reported outcomes are assessed at 3 months postoperatively
  Interventions: Device: Extended Depth of Focus Intraocular Lens Implantation

INTERVENTIONS:
Device: Extended Depth of Focus Intraocular Lens Implantation — Bilateral implantation of the AcrySof IQ Vivity (Alcon, Fort Worth, TX, USA) Extended Depth of Focus (EDOF) intraocular lens during phacoemulsification cataract surgery. The Vivity is a single-piece hydrophobic acrylic IOL (6.0 mm optic, 13.0 mm overall length) featuring non-diffractive X-WAVE wavefront-shaping technology with a slightly elevated central plateau (~1 µm) and surrounding curvature modulation to extend focal range. It incorporates UV and blue light filtering with refractive index 1.55 at 35°C. The spherical model (powers +15.0 D to +25.0 D) or toric model (cylinder 1.03 D to 4.11 D at IOL plane) is selected based on corneal astigmatism. IOL power calculated using Kane formula targeting emmetropia. Surgery performed with 2.2 mm incision under topical anesthesia, with second-eye surgery within 7 days. This study specifically evaluates performance in patients with early-stage stable keratoconus.

SUMMARY:
The goal of this clinical trial is to learn if the Vivity Extended Depth of Focus intraocular lens works to improve vision in adults with cataracts and early-stage keratoconus. It will also learn about the safety and tolerance of this premium lens in patients with mild corneal irregularities. The main questions it aims to answer are:

* Does the Vivity EDOF lens provide good distance vision (20/25 or better) in the dominant eye at 3 months after surgery?
* Does it improve vision at intermediate and near distances compared to before surgery?
* Does it preserve contrast sensitivity and optical quality despite mild corneal irregularities?
* What is the patient-reported quality of life and satisfaction after implantation?
* What visual disturbances (such as halos) do participants experience?

All participants will:

* Receive the Vivity EDOF intraocular lens (or its toric version if astigmatism is present) in both eyes during standard cataract surgery, with the second eye operated within 7 days;
* Undergo comprehensive eye examinations before surgery including vision testing, corneal imaging, and optical quality measurements;
* Attend a follow-up visit at 3 months after surgery for detailed vision testing at multiple distances, contrast sensitivity testing under different lighting conditions, halo assessment, and quality-of-life questionnaires.

DETAILED DESCRIPTION:
Background and Rationale Keratoconus (KC) is a progressive, non-inflammatory corneal ectasia characterized by stromal thinning and irregular astigmatism, often resulting in significant higher-order aberrations (HOAs) that impair visual quality. Due to these optical limitations, the use of premium intraocular lenses (pIOLs) has traditionally been considered contraindicated in these patients. However, in patients with early-stage keratoconus, corneal shape and optical quality can be relatively well preserved, with HOAs remaining within acceptable limits. These patients may thus benefit from carefully selected premium IOL technologies.

Extended-depth-of-focus (EDOF) IOLs, in contrast to traditional multifocal lenses, not only provide significantly fewer visual disturbances but, thanks to their elongated focus, they could mitigate HOAs and coma-like distortions characteristic of early keratoconus. Unlike monofocal or multifocal lenses, which rely on a single, sharp focal point or discrete focal planes, EDOF lenses are inherently designed to maintain functional retinal image quality across an extended focal range, offering greater tolerance to minor defocus and wavefront aberrations. While EDOF lenses do not correct such aberrations, their extended focal range may reduce the impact of this distortion on functional vision. This is especially true for non-diffractive EDOF lenses, which preserve high levels of contrast sensitivity by not splitting light energy into multiple focal points.

The AcrySof IQ Vivity IOL (Alcon, Fort Worth, TX, USA) is a non-diffractive EDOF IOL that uses wavefront-shaping technology to elongate the focal range. Previous studies have already demonstrated good outcomes in patients with other challenging ocular conditions such as glaucoma, macular degeneration, and epiretinal membrane. The present pilot study aims to evaluate the visual performance, tolerance, and optical quality outcomes following implantation of the Vivity IOL in patients with cataract and stable, early-stage keratoconus. This investigation explores the clinical viability of premium IOLs in a population traditionally excluded from such refractive options.

Study Design This is a prospective, interventional, single-center pilot study conducted in Italy. The study has been approved by the local ethics committee (protocol number 22546) and adheres to the principles of the Declaration of Helsinki. A total of 10 patients (20 eyes) with cataracts and mild bilateral keratoconus will be enrolled and followed for 3 months after bilateral implantation of the AcrySof IQ Vivity EDOF IOL.

Study Objectives

Primary Objective:

- To evaluate monocular distance-corrected visual acuity (DCVA) in the dominant eye at 3 months after surgery.

Secondary Objectives:

* To assess monocular and binocular uncorrected and distance-corrected visual acuity at distance (4 meters), intermediate (66 cm), and near (40 cm)
* To evaluate binocular defocus curves from +1.50 D to -3.50 D in 0.50 D increments;
* To measure monocular and binocular contrast sensitivity under photopic (80 cd/m²), mesopic (6 cd/m²), and scotopic (3 cd/m²) lighting conditions;
* To assess ocular optical quality including root mean square (RMS) wavefront error and point spread function (PSF) Strehl ratio at 3 mm and 4 mm pupil diameters;
* To evaluate binocular halo perception using standardized halometry;
* To assess patient-reported quality of life using the National Eye Institute Refractive Error Quality of Life Instrument-42 (NEI-RQL-42) questionnaire;
* To evaluate the safety profile including intra- and postoperative complications and adverse events;
* To assess toric IOL rotational stability in eyes receiving the toric version.

Eligibility criteria such as inclusion and exclusion criteria are reported separately.

Preoperative Assessment:

All patients will receive a comprehensive ophthalmologic evaluation prior to surgery, including:

* Measurement of monocular and binocular uncorrected and corrected visual acuity for distance (4 meters) and near (40 cm) using CSO Vision Charts software version 14.0
* Corneal tomography using MS-39 anterior segment optical coherence tomography (CSO, Florence, Italy)
* Ocular optical quality analysis using Pyramidal WaveFront-based sensor aberrometer (Osiris T Aberrometer, CSO, Florence, Italy) to assess higher-order aberrations including coma and coma-like aberrations
* Optical biometry using Lenstar 900 (Haag-Streit Diagnostics, Koeniz, Switzerland) for axial length and IOL power calculation
* Intraocular pressure measurement
* Slit-lamp examination of the anterior segment
* Dilated fundoscopy
* Macular evaluation through spectral-domain optical coherence tomography (Spectralis OCT, Heidelberg Engineering GmbH, Germany)
* Ocular dominance determination using the Miles test

Surgical Procedure:

All patients will undergo standard phacoemulsification cataract surgery performed by the same experienced surgeon using a 2.2 mm phaco probe under topical anesthesia. The AcrySof IQ Vivity EDOF IOL will be implanted in the capsular bag with a target of emmetropia bilaterally. IOL power calculation will be performed using the Kane formula. In eyes with regular corneal astigmatism equal to or greater than 1.00 diopter, the toric version of the Vivity IOL (AcrySof IQ Vivity Toric) will be implanted to optimize postoperative refractive outcomes. The second eye will be operated within 7 days of the first eye surgery.

Postoperative Follow-up:

Toric IOL rotational stability will be assessed on postoperative days 1 and 7 to account for early positional shifts and to allow for re-centering if necessary. The IOL will be deemed stable if the angular deviation is less than 5 degrees and if it induces a residual cylindrical error of 0.75 diopters or less, as estimated using the Toric IOL Assistant feature of the Osiris T Aberrometer.

Complete ophthalmological examination will be performed at the 3-month follow-up visit and outcome measures are measured as explained in the outcome measures section.

The Vivity IOL Technology The AcrySof IQ Vivity is a single-piece, hydrophobic acrylic EDOF IOL that utilizes a non-diffractive wavefront-shaping mechanism to enhance intermediate and near vision. The optic is 6.0 mm in diameter with an overall length of 13.0 mm and features a C-loop haptic design. The lens material incorporates both ultraviolet and blue light-filtering chromophores and has a refractive index of 1.55 at 35°C.

The lens design is based on a monofocal aspheric platform with an aberration-neutral anterior surface. The central optical zone incorporates X-WAVE technology, which integrates two subtle anterior surface transition elements: a slightly elevated central plateau (approximately 1 micrometer) that stretches the wavefront to extend the focus, and a surrounding curvature modulation that shifts the wavefront, ensuring efficient retinal energy delivery across the extended range.

The spherical model is available in powers ranging from +15.0 diopters to +25.0 diopters in 0.5 diopter increments, with additional availability up to +30.0 diopters in selected markets. The toric version, AcrySof IQ Vivity Toric, incorporates the same non-diffractive EDOF design and is offered in cylinder powers from 1.03 diopters to 4.11 diopters at the IOL plane.

Statistical Analysis All statistical analyses will be performed using STATA software, version 13.0 (StataCorp, College Station, TX, USA). The distribution of continuous variables will be assessed with the Shapiro-Wilk test. When data are normally distributed, results will be reported as mean ± standard deviation.

To evaluate the safety profile of the implanted IOL, both absolute and relative frequencies of intra- and postoperative complications, as well as any adverse events, will be recorded and analyzed at each follow-up. Paired t-tests will be conducted between preoperative and postoperative DCVA, DCNVA, UDVA, UNVA, and total RMS to assess postoperative functional improvement.

The primary endpoint is the evaluation of DCVA in the dominant eye at 3 months. A formal sample-size calculation was performed based on a previous pilot series reporting a standard deviation of 0.01 logMAR for monocular DCVA in eyes with stable keratoconus and cataract implanted with a premium IOL. A single-group design was used to estimate a 95% confidence interval for one standard deviation via the chi-square method. Assuming a standard deviation of 0.017 logMAR, 10 subjects (10 eyes) are required to yield a confidence interval half-width no greater than 0.02 logMAR (equivalent to one ETDRS letter). Sample-size calculations were carried out with PASS 2023, version 23.0.2.

Safety Considerations All participants will be carefully monitored for any adverse events or complications related to the surgical procedure or the implanted IOL. Standard cataract surgery risks include infection (endophthalmitis), inflammation, bleeding, increased intraocular pressure, lens dislocation, posterior capsule rupture, cystoid macular edema, and retinal detachment. Additional considerations specific to premium IOLs include the potential for visual disturbances such as glare, halos, starbursts, reduced contrast sensitivity, and in rare cases, dissatisfaction requiring IOL exchange.

In the specific context of keratoconus patients, there is theoretical concern that residual corneal irregularities and higher-order aberrations might interact with the IOL optics in unpredictable ways, potentially limiting visual quality or increasing photic phenomena. However, by carefully selecting only patients with early-stage, stable keratoconus and relatively preserved corneal morphology, this study aims to minimize these risks while exploring the potential benefits of EDOF technology in this population.

Any serious adverse events will be immediately reported to the ethics committee and appropriate medical management will be provided. Participants are free to withdraw from the study at any time without affecting their medical care.

Expected Outcomes and Significance This pilot study will provide preliminary evidence regarding the safety, efficacy, and patient satisfaction associated with Vivity EDOF IOL implantation in patients with early-stage keratoconus. If successful, the results may challenge the traditional view that premium IOLs are contraindicated in keratoconus and open new treatment options for carefully selected patients who wish to reduce spectacle dependence after cataract surgery.

The non-diffractive EDOF design of the Vivity lens, with its extended focal range and preserved contrast sensitivity, may be particularly well-suited to tolerating the mild corneal irregularities present in early keratoconus. By extending the depth of focus rather than creating discrete focal points, the lens may maintain functional vision despite minor wavefront aberrations.

Results from this study will inform larger, multicenter, randomized controlled trials and may ultimately contribute to updated clinical guidelines for IOL selection in keratoconus patients

ELIGIBILITY:
Inclusion Criteria:

* Adults requiring bilateral cataract surgery
* Mild bilateral keratoconus defined as stage 0-1 according to the ABCD classification system
* Keratoconus stability defined as maximum keratometry (K) changes less than 1 diopter and maximum pachymetry reduction less than 2% within the previous 5 years
* Pre-cataract spectacle distance-corrected visual acuity of 0.1 to 0.0 LogMAR (Snellen 20/25 to 20/20)
* Agreement to bilateral implantation of AcrySof IQ Vivity Extended Depth of Focus intraocular lens
* Willingness to undergo second-eye surgery within 7 days after first-eye procedure
* Ability and willingness to attend all scheduled follow-up visits as per study protocol
* Provision of written informed consent to participate in the study

Exclusion Criteria:

* Any ocular comorbidities other than cataract and keratoconus, or history of any disease that could affect visual results (e.g., glaucoma, retinal disorders)
* Corneal opacity including any corneal scarring
* Advanced or progressive keratoconus
* Any previous ocular surgery other than corneal cross-linking performed at least 5 years prior to enrollment
* Corneal cross-linking performed within 5 years prior to enrollment
* Amblyopia
* Pseudoexfoliation syndrome or zonular laxity
* History of uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Distance-Corrected Visual Acuity in the Dominant Eye | 3 months after surgery
  Monocular distance-corrected visual acuity (DCVA) measured in the dominant eye at 4 meters using CSO Vision Charts software version 14.0, recorded in logMAR units. Lower logMAR values indicate better visual acuity (e.g., 0.0 logMAR = Snellen 20/20; 0.1 logMAR = Snellen 20/25). Visual acuity is measured with best spectacle correction to assess the maximum visual performance achievable with the implanted IOL. The target outcome is DCVA of 0.1 logMAR (20/25) or better, indicating clinically excellent visual function. This primary endpoint evaluates whether the Vivity EDOF IOL can maintain high-quality distance vision despite the presence of mild corneal irregularities characteristic of early keratoconus

SECONDARY OUTCOMES:
Monocular and Binocular Uncorrected Distance Visual Acuity | Baseline (preoperative) and 3 months after surgery
  Uncorrected distance visual acuity (UDVA) measured at 4 meters without spectacles using CSO Vision Charts version 14.0, recorded in logMAR units for each eye separately (monocular) and both eyes together (binocular). Lower logMAR values indicate better visual acuity. This outcome assesses spectacle independence for distance vision tasks such as driving and watching television. Results will be compared to preoperative values to determine visual improvement.
Monocular and Binocular Uncorrected and Distance-Corrected Near Visual Acuity | Baseline (preoperative) and 3 months after surgery
  Near visual acuity measured at 40 cm both without spectacles (UNVA) and with distance correction (DCNVA), using CSO Vision Charts version 14.0, recorded in logMAR units monocularly and binocularly. Lower logMAR values indicate better near vision. This outcome evaluates the EDOF lens's ability to provide functional near vision for reading and smartphone use, both with and without glasses, assessing spectacle independence for near tasks. Results will be compared to preoperative values
Monocular and Binocular Uncorrected and Distance-Corrected Intermediate Visual Acuity | 3 months after surgery
  Intermediate visual acuity measured at 66 cm both without spectacles (UI66VA) and with distance correction (DCI66VA), using CSO Vision Charts version 14.0, recorded in logMAR units monocularly and binocularly. Lower logMAR values indicate better intermediate vision. This outcome evaluates functional vision for computer work, dashboard viewing, and other arm's-length tasks, which is a key advantage of EDOF IOLs, both with and without spectacle correction.
Binocular Defocus Curve Visual Acuity Profile | 3 months after surgery
  Visual acuity measured binocularly across a range of defocus from +1.50 diopters to -3.50 diopters in 0.50 diopter increments, relative to best distance correction, using CSO Vision Charts version 14.0 with randomized letter sequences. Results plotted as logMAR visual acuity versus defocus level; lower logMAR values at each defocus level indicate better performance. This outcome characterizes the continuous range of functional vision provided by the EDOF lens from distance through intermediate to near. Positive defocus simulates hyperopia (distance blur); negative defocus simulates near viewing distances.
Monocular and Binocular Contrast Sensitivity Under Photopic, Mesopic, and Scotopic Conditions | 3 months after surgery
  Contrast sensitivity measured monocularly and binocularly at multiple spatial frequencies (3, 6, 12, and 18 cycles per degree) under three lighting conditions using CSV-1000 HGT testing (Vector Vision, Greenville, OH), recorded in log units: photopic (bright light, 80 cd/m²), mesopic (dim light, 6 cd/m²), and scotopic (dark-adapted, 3 cd/m²). Higher log values indicate better contrast sensitivity. This outcome evaluates the ability to detect contrast and fine detail across different lighting environments, bright daylight, twilight/indoor low-light, and nighttime conditions, which is critical for reading, face recognition, driving, and overall visual quality. Contrast sensitivity under reduced lighting is often compromised with multifocal IOLs but may be preserved with non-diffractive EDOF designs.
Total Root Mean Square (RMS) Wavefront Error | 3 months after surgery
  Total ocular higher-order aberrations measured using Pyramidal WaveFront-based aberrometer (Osiris T Aberrometer, CSO, Florence, Italy), recorded as RMS in micrometers. Lower RMS values indicate better optical quality with fewer aberrations. This objective measure evaluates whether the IOL implantation reduces the overall optical irregularities present preoperatively in keratoconus eyes. Results will be compared between preoperative and postoperative measurements
Root Mean Square Wavefront Error at 3 mm and 4 mm Pupil Diameters | 3 months after surgery
  Root mean square (RMS) wavefront error measured at both 3 mm and 4 mm pupil diameters using Osiris T Aberrometer, recorded in micrometers. Lower RMS values indicate fewer optical aberrations and better optical quality. These metrics characterize optical performance under photopic conditions (3 mm pupil, naturally constricted) and mesopic conditions (4 mm pupil, moderate dilation), which may reveal greater interaction between corneal irregularities and IOL optics as pupil size increases.
Point Spread Function Strehl Ratio at 3 mm and 4 mm Pupil Diameters | 3 months after surgery
  Point spread function (PSF) Strehl ratio measured at both 3 mm and 4 mm pupil diameters using Osiris T Aberrometer. The Strehl ratio ranges from 0 to 1, with higher values indicating better retinal image quality and values closer to 1.0 representing diffraction-limited optical performance. These metrics quantify how efficiently light is focused onto the retina under photopic (3 mm pupil) and mesopic (4 mm pupil) conditions, providing objective assessment of functional optical quality in keratoconus eyes with EDOF IOLs.
Binocular Halo Perception Using Aston Halometer | 3 months after surgery
  Subjective halo size and intensity measured binocularly using the Aston Halometer, which displays a standardized central LED glare source (5000 K) on an iPad4. Participants indicate the perceived halo size on a radial scale. Smaller halo measurements indicate less photic disturbance. This outcome assesses one of the most common visual complaints with premium IOLs, particularly relevant for night driving and assessing tolerance in keratoconus eyes with residual aberrations.
NEI-RQL-42 Quality of Life Scores | 3 months after surgery
  Patient-reported quality of life measured using the National Eye Institute Refractive Error Quality of Life Instrument-42 (NEI-RQL-42) questionnaire, consisting of 13 subscales with 42 items across 16 question/response formats. Each item is converted to a 0-100 scale, with higher scores indicating better vision-related quality of life. Subscales include clarity of vision, expectations, near vision, far vision, diurnal fluctuations, activity limitations, glare, symptoms, dependence on correction, worry, suboptimal correction, appearance, and satisfaction with correction. This validated instrument captures patient-centered functional outcomes and satisfaction.
Incidence of Intraoperative and Postoperative Adverse Events | From surgery through 3 months postoperatively
  All intraoperative complications (e.g., posterior capsule rupture, zonular dehiscence, vitreous loss) and postoperative adverse events (e.g., endophthalmitis, increased intraocular pressure, cystoid macular edema, retinal detachment, persistent inflammation, IOL dislocation) recorded as absolute and relative frequencies. This outcome evaluates the safety profile of premium IOL implantation specifically in the keratoconus population. Lower frequencies indicate better safety.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Integrata di Verona, Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farideh D, Azad S, Feizollah N, Sana N, Cyrus A, Mohammad G, Alireza BR. Clinical outcomes of new toric trifocal diffractive intraocular lens in patients with cataract and stable keratoconus: Six months follow-up. Medicine (Baltimore). 2017 Mar;96(12):e6340. doi: 10.1097/MD.0000000000006340. PMID 28328814
- [Background] Rampat R, Gatinel D. Multifocal and Extended Depth-of-Focus Intraocular Lenses in 2020. Ophthalmology. 2021 Nov;128(11):e164-e185. doi: 10.1016/j.ophtha.2020.09.026. Epub 2020 Sep 25. PMID 32980397
- [Background] Pedrotti E, Chierego C, Talli PM, Selvi F, Galzignato A, Neri E, Barosco G, Montresor A, Rodella A, Marchini G. Extended Depth of Focus Versus Monofocal IOLs: Objective and Subjective Visual Outcomes. J Refract Surg. 2020 Apr 1;36(4):214-222. doi: 10.3928/1081597X-20200212-01. PMID 32267951
- [Background] Palomino-Bautista C, Sanchez-Jean R, Carmona-Gonzalez D, Pinero DP, Molina-Martin A. Subjective and objective depth of field measures in pseudophakic eyes: comparison between extended depth of focus, trifocal and bifocal intraocular lenses. Int Ophthalmol. 2020 Feb;40(2):351-359. doi: 10.1007/s10792-019-01186-6. Epub 2019 Oct 3. PMID 31583551
- [Background] Gillmann K, Mermoud A. Visual Performance, Subjective Satisfaction and Quality of Life Effect of a New Refractive Intraocular Lens with Central Extended Depth of Focus. Klin Monbl Augenheilkd. 2019 Apr;236(4):384-390. doi: 10.1055/a-0799-9700. Epub 2019 Feb 14. PMID 30763956
- [Background] Pedrotti E, Mastropasqua R, Passilongo M, Parisi G, Marchesoni I, Marchini G. Comparison of two multifocal intraocular lens designs that differ only in near add. J Refract Surg. 2014 Nov;30(11):754-60. doi: 10.3928/1081597X-20141021-07. PMID 25375848
- [Background] Alio JL, Pinero DP, Plaza-Puche AB, Amparo F, Jimenez R, Rodriguez-Prats JL, Javaloy J. Visual and optical performance with two different diffractive multifocal intraocular lenses compared to a monofocal lens. J Refract Surg. 2011 Aug;27(8):570-81. doi: 10.3928/1081597X-20101223-01. Epub 2011 Jan 3. PMID 21210572
- [Background] Gil MA, Varon C, Cardona G, Vega F, Buil JA. Comparison of far and near contrast sensitivity in patients symmetrically implanted with multifocal and monofocal IOLs. Eur J Ophthalmol. 2014 Jan-Feb;24(1):44-52. doi: 10.5301/ejo.5000335. Epub 2013 Jun 24. PMID 23813113
- [Background] Buckhurst PJ, Naroo SA, Davies LN, Shah S, Drew T, Wolffsohn JS. Assessment of dysphotopsia in pseudophakic subjects with multifocal intraocular lenses. BMJ Open Ophthalmol. 2017 Jun 19;1(1):e000064. doi: 10.1136/bmjophth-2016-000064. eCollection 2017. PMID 29354708
- [Background] de Silva SR, Evans JR, Kirthi V, Ziaei M, Leyland M. Multifocal versus monofocal intraocular lenses after cataract extraction. Cochrane Database Syst Rev. 2016 Dec 12;12(12):CD003169. doi: 10.1002/14651858.CD003169.pub4. PMID 27943250
- [Background] Flockerzi E, Vinciguerra R, Belin MW, Vinciguerra P, Ambrosio R Jr, Seitz B. Combined biomechanical and tomographic keratoconus staging: Adding a biomechanical parameter to the ABCD keratoconus staging system. Acta Ophthalmol. 2022 Aug;100(5):e1135-e1142. doi: 10.1111/aos.15044. Epub 2021 Oct 16. PMID 34655452
- [Background] Vandevenne MMS, Webers VSC, Segers MHM, Berendschot TTJM, Zadok D, Dickman MM, Nuijts RMMA, Abulafia A. Accuracy of intraocular lens calculations in eyes with keratoconus. J Cataract Refract Surg. 2023 Mar 1;49(3):229-233. doi: 10.1097/j.jcrs.0000000000001088. Epub 2022 Oct 28. PMID 36314969
- [Background] Haigis W. Challenges and approaches in modern biometry and IOL calculation. Saudi J Ophthalmol. 2012 Jan;26(1):7-12. doi: 10.1016/j.sjopt.2011.11.007. PMID 23960962
- [Background] Hashemi H, Heydarian S, Hooshmand E, Saatchi M, Yekta A, Aghamirsalim M, Valadkhan M, Mortazavi M, Hashemi A, Khabazkhoob M. The Prevalence and Risk Factors for Keratoconus: A Systematic Review and Meta-Analysis. Cornea. 2020 Feb;39(2):263-270. doi: 10.1097/ICO.0000000000002150. PMID 31498247